CLINICAL TRIAL: NCT06334666
Title: The Efficacy of Pedometer-motivated Physical Activity for the Management of Patients With Metabolic-associated Steatotic Liver Disease: a Randomized-controlled Trial
Brief Title: The Efficacy of Pedometer-motivated Physical Activity for the Management of Patients With MASLD.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI 172/2024
Record Dates: First submitted 2024-03-18; First posted 2024-03-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Daily Step Count; MASLD; BMI; Metabolic Syndrome; NAFLD; Insulin Resistance; Genetic Polymorphism; Cardiovascular Disease (CVD)
Keywords: Daily step count; MASLD; Pedometer; BMI; Metabolic Syndrome; NAFLD; Insulin Resistance; Genetic polymorphism; Cardiovascular disease (CVD)
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Insulin Resistance; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Encourage using pedometer group. (Experimental): MASLD patient who received pedometer recording and was encouraged to use actively.
  Interventions: Other: Encourage using pedometer
- Placebo comparator: Discourage using pedometer group (No Intervention): MASLD patient who received pedometer recording but without encouraged to use.

INTERVENTIONS:
Other: Encourage using pedometer — MASLD patient used pedometer recording actively with encourage by care provider or investigator
  Arms: Active Comparator: Encourage using pedometer group.

SUMMARY:
The study conducted a health survey among Thai adults in 2022 and found a significant increase in obesity and nonalcoholic fatty liver disease (NAFLD), leading to metabolic-associated steatotic liver disease (MASLD). The prevalence of NAFLD was 19.7%, with higher rates in individuals with metabolic syndrome and diabetes. MASLD is associated with insulin resistance and genetic polymorphisms, particularly the patatin like phospholipase domain containing 3-rs738409 variant. Additionally, physical activity was inversely related to liver disease risk, with higher step counts associated with reduced incidence of NAFLD and liver-related mortality. The study aims to investigate the impact of dietary advice and pedometer use on physical activity levels and health outcomes in MASLD patients over 24 weeks.

DETAILED DESCRIPTION:
The results of the health survey of the Thai population through physical examinations in the year 2022 found that among Thai people aged 18 and older, the prevalence of obesity (BMI ≥25 kg/m2) was 44.9% (40.3% in males and 49.2% in females), which has increased significantly over the past decades. This condition is a significant factor contributing to the rising incidence of nonalcoholic fatty liver disease (NAFLD) among the Thai population. NAFLD refers to fatty liver disease in individuals who consume alcohol in amounts less than 140 grams per week for females or less than 210 grams per week for males. Those with clinical features of metabolic dysfunction have been newly defined as having metabolic-associated steatotic liver disease (MASLD).

In this survey of 18,588 individuals, the prevalence of NAFLD was 19.7%, with rates of 20.9% in males and 18.6% in females. It was notably higher at 43.5% in individuals with abdominal obesity (metabolic syndrome) and 35.6% in individuals with diabetes. Factors such as age, sex, physical activity, smoking, and metabolic characteristics such as overweight or obesity, abdominal obesity, high triglyceride levels, diabetes, hypertension, and low HDL cholesterol levels are significantly associated with NAFLD.

MASLD, a type of fatty liver disease, is directly associated with insulin resistance, a key risk factor for cardiovascular diseases. Current treatment guidelines for MASLD have clear evidence that weight loss through dietary control and appropriate physical activity or exercise can reduce fat accumulation in the liver, inflammation, and fibrosis. Importantly, it also improves various metabolic parameters such as blood sugar and lipid levels, as well as the effectiveness of insulin.

The etiology of MASLD is related to behavioral and environmental factors, such as high-calorie diets combined with low physical activity and sedentary lifestyles. These factors promote insulin resistance, stimulating lipolysis and the movement of free fatty acids to various organs, including the liver. This leads to fat accumulation in the liver, insulin-resistant hepatic tissue, abnormal β-oxidation processes, oxidative stress, hepatic inflammation, increased stellate cell activation, and subsequent fibrosis, eventually increasing the risk of liver cirrhosis and hepatocellular carcinoma.

Genetic polymorphisms play a significant role in MASLD pathogenesis, with single nucleotide polymorphisms (SNPs) in the patatin like phospholipase domain containing-3 gene, particularly the rs738409 variant, being strongly associated with fat accumulation and fibrosis in the liver.

Furthermore, a systematic review and analysis of data from 12 studies involving 111,309 individuals found that the number of steps per day, particularly 8,800 steps per day, was associated with a significant reduction in the risk of overall mortality and cardiovascular diseases (CVD). Additionally, increasing physical activity was associated with a reduced risk of chronic liver disease overall and NAFLD specifically. Increasing physical activity by 2,500 steps per day was associated with a 38% reduction in chronic liver disease and a 47% reduction in NAFLD, regardless of obesity status.

This research aims to conduct a randomized study to provide advice to MASLD patients to modify their diet and wear pedometers to encourage changes in physical activity, with a goal of achieving at least 8,800 steps per day, compared to MASLD patients who only receive dietary advice and wear pedometers to record daily steps over a 24-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be diagnosed with MASLD according to the diagnostic criteria of the A multi-society Delphi consensus statement on new fatty liver disease nomenclature 2023, with evidence of hepatic steatosis and alcohol consumption of less than 140 grams per week for females or less than 210 grams per week for males, along with at least one of the clinical characteristics of metabolic syndrome.
2. Participants must be at least 18 years old at the time of enrollment.
3. Patients must consent to blood testing for the identification of the patatin like phospholipase domain containing-3 gene polymorphism.

Exclusion Criteria:

1. Individuals who engage in regular exercise for at least 20 minutes per day, at least 3 days per week.
2. Individuals who have regular physical activity with walking exceeding 3000 steps per day before participating in the study.
3. Individuals diagnosed with other chronic liver diseases such as hepatitis B or C, autoimmune hepatitis, Wilson's disease, liver cancer, hemochromatosis, liver cirrhosis, or others.
4. Individuals diagnosed with diseases that may affect non-alcoholic fatty liver disease, such as HIV, various chronic inflammatory diseases, or connective tissue disorders.
5. Individuals taking medications known to promote fatty liver disease, including amiodarone, steroids, methotrexate, hormonal medications, or immunosuppressants.
6. Individuals who have previously taken medications known to impact fatty liver disease, including vitamin E, pioglitazone, Glucagon-like peptide-1 agonists, SGLT2 inhibitors.
7. Participants intending to join weight loss programs or undergo bariatric surgery for obesity treatment.
8. Individuals with cirrhosis.
9. Individuals diagnosed with liver cancer.
10. Individuals with severe chronic diseases still exhibiting symptoms during physical activity that may exacerbate the disease, such as coronary artery disease, chronic obstructive pulmonary disease, or severe osteoarthritis.
11. Patients with contraindications for undergoing MRI examinations, such as claustrophobia or having body implants or materials that are incompatible with MRI scanning.
12. Women who are pregnant.
13. Individuals who do not provide formal consent to participate in the research project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To compare the changes in hepatic fat accumulation assessed by MRI-PDFF between the MASLD patient group wearing pedometers to promote physical activity, compared to the MASLD patient group with normal daily walking behavior. | 24 weeks
  To compare the changes in hepatic fat accumulation assessed by magnetic resonance imaging proton-density fat fraction (MRI-PDFF) between the MASLD patient group wearing pedometers to promote achieving at least 8,800 steps per day, compared to the MASLD patient group with normal daily walking behavior, along with dietary adjustments.

SECONDARY OUTCOMES:
To compare changes in metabolic parameters between the MASLD patient group wearing pedometers to promote physical activity, compared to the MASLD patient group with normal daily walking behavior, along with dietary adjustments. | 24 weeks
  To compare changes in various metabolic parameters(e.g. weight in kilograms, height in meters, blood sugar levels such as FBS in milligrams per deciliter or HbA1C in percentage , and blood lipid profiles such as total cholesteral in milligrams per deciliter) between the MASLD patient group wearing pedometers to promote achieving at least 8,800 steps per day, compared to the MASLD patient group with normal daily walking behavior, along with dietary adjustments.
To study the impact of genes on changes in hepatic fat accumulation between the MASLD patient group wearing pedometers to promote physical activity, compared to the MASLD patient group with normal daily walking behavior. | 24 weeks
  To study the impact of the patatin like phospholipase domain containing-3 rs738409 G alleles on changes in hepatic fat accumulation assessed by MRI-PDFF between the MASLD patient group wearing pedometers to promote achieving at least 8,800 steps per day, compared to the MASLD patient group with normal daily walking behavior, along with dietary adjustments.

CONTACTS AND LOCATIONS:
Overall Officials: Division of Gastroenterology, Siriraj Hospital, Principal Investigator — Siriraj Hospital; Phunchai Charatcharoenwitthaya, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Result] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Result] Ekstedt M, Nasr P, Kechagias S. Natural History of NAFLD/NASH. Curr Hepatol Rep. 2017;16(4):391-397. doi: 10.1007/s11901-017-0378-2. Epub 2017 Nov 13. PMID 29984130
- [Result] Engin A. The Definition and Prevalence of Obesity and Metabolic Syndrome. Adv Exp Med Biol. 2017;960:1-17. doi: 10.1007/978-3-319-48382-5_1. PMID 28585193
- [Result] Goodpaster BH, Katsiaras A, Kelley DE. Enhanced fat oxidation through physical activity is associated with improvements in insulin sensitivity in obesity. Diabetes. 2003 Sep;52(9):2191-7. doi: 10.2337/diabetes.52.9.2191. PMID 12941756
- [Result] Jeon CY, Lokken RP, Hu FB, van Dam RM. Physical activity of moderate intensity and risk of type 2 diabetes: a systematic review. Diabetes Care. 2007 Mar;30(3):744-52. doi: 10.2337/dc06-1842. PMID 17327354
- [Result] White T, Westgate K, Wareham NJ, Brage S. Estimation of Physical Activity Energy Expenditure during Free-Living from Wrist Accelerometry in UK Adults. PLoS One. 2016 Dec 9;11(12):e0167472. doi: 10.1371/journal.pone.0167472. eCollection 2016. PMID 27936024
- [Result] LaMonte MJ, Lewis CE, Buchner DM, Evenson KR, Rillamas-Sun E, Di C, Lee IM, Bellettiere J, Stefanick ML, Eaton CB, Howard BV, Bird C, LaCroix AZ. Both Light Intensity and Moderate-to-Vigorous Physical Activity Measured by Accelerometry Are Favorably Associated With Cardiometabolic Risk Factors in Older Women: The Objective Physical Activity and Cardiovascular Health (OPACH) Study. J Am Heart Assoc. 2017 Oct 17;6(10):e007064. doi: 10.1161/JAHA.117.007064. PMID 29042429
- [Result] Kim D, Murag S, Cholankeril G, Cheung A, Harrison SA, Younossi ZM, Ahmed A. Physical Activity, Measured Objectively, Is Associated With Lower Mortality in Patients With Nonalcoholic Fatty Liver Disease. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1240-1247.e5. doi: 10.1016/j.cgh.2020.07.023. Epub 2020 Jul 16. PMID 32683103
- [Result] Saint-Maurice PF, Troiano RP, Berrigan D, Kraus WE, Matthews CE. Volume of Light Versus Moderate-to-Vigorous Physical Activity: Similar Benefits for All-Cause Mortality? J Am Heart Assoc. 2018 Apr 2;7(7):e008815. doi: 10.1161/JAHA.118.008815. PMID 29610219
- [Result] Bird SR, Hawley JA. Update on the effects of physical activity on insulin sensitivity in humans. BMJ Open Sport Exerc Med. 2017 Mar 1;2(1):e000143. doi: 10.1136/bmjsem-2016-000143. eCollection 2016. PMID 28879026
- [Result] Kwak MS, Kim D, Chung GE, Kim W, Kim JS. The preventive effect of sustained physical activity on incident nonalcoholic fatty liver disease. Liver Int. 2017 Jun;37(6):919-926. doi: 10.1111/liv.13332. Epub 2016 Dec 24. PMID 27917585
- [Result] Kistler KD, Brunt EM, Clark JM, Diehl AM, Sallis JF, Schwimmer JB; NASH CRN Research Group. Physical activity recommendations, exercise intensity, and histological severity of nonalcoholic fatty liver disease. Am J Gastroenterol. 2011 Mar;106(3):460-8; quiz 469. doi: 10.1038/ajg.2010.488. Epub 2011 Jan 4. PMID 21206486
- [Result] Asada F, Nomura T, Hosui A, Kubota M. Influence of increased physical activity without body weight loss on hepatic inflammation in patients with nonalcoholic fatty liver disease. Environ Health Prev Med. 2020 Jun 10;25(1):18. doi: 10.1186/s12199-020-00857-6. PMID 32522147
- [Result] Karlas T, Petroff D, Sasso M, Fan JG, Mi YQ, de Ledinghen V, Kumar M, Lupsor-Platon M, Han KH, Cardoso AC, Ferraioli G, Chan WK, Wong VW, Myers RP, Chayama K, Friedrich-Rust M, Beaugrand M, Shen F, Hiriart JB, Sarin SK, Badea R, Jung KS, Marcellin P, Filice C, Mahadeva S, Wong GL, Crotty P, Masaki K, Bojunga J, Bedossa P, Keim V, Wiegand J. Individual patient data meta-analysis of controlled attenuation parameter (CAP) technology for assessing steatosis. J Hepatol. 2017 May;66(5):1022-1030. doi: 10.1016/j.jhep.2016.12.022. Epub 2016 Dec 28. PMID 28039099
- [Result] Stine JG, Munaganuru N, Barnard A, Wang JL, Kaulback K, Argo CK, Singh S, Fowler KJ, Sirlin CB, Loomba R. Change in MRI-PDFF and Histologic Response in Patients With Nonalcoholic Steatohepatitis: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2274-2283.e5. doi: 10.1016/j.cgh.2020.08.061. Epub 2020 Aug 31. PMID 32882428
- [Result] Hernaez R, Lazo M, Bonekamp S, Kamel I, Brancati FL, Guallar E, Clark JM. Diagnostic accuracy and reliability of ultrasonography for the detection of fatty liver: a meta-analysis. Hepatology. 2011 Sep 2;54(3):1082-1090. doi: 10.1002/hep.24452. PMID 21618575
- [Result] Shen J, Wong GL, Chan HL, Chan RS, Chan HY, Chu WC, Cheung BH, Yeung DK, Li LS, Sea MM, Woo J, Wong VW. PNPLA3 gene polymorphism and response to lifestyle modification in patients with nonalcoholic fatty liver disease. J Gastroenterol Hepatol. 2015 Jan;30(1):139-46. doi: 10.1111/jgh.12656. PMID 25040896
- [Result] Romero-Gomez M, Zelber-Sagi S, Trenell M. Treatment of NAFLD with diet, physical activity and exercise. J Hepatol. 2017 Oct;67(4):829-846. doi: 10.1016/j.jhep.2017.05.016. Epub 2017 May 23. PMID 28545937
- [Result] Koutoukidis DA, Koshiaris C, Henry JA, Noreik M, Morris E, Manoharan I, Tudor K, Bodenham E, Dunnigan A, Jebb SA, Aveyard P. The effect of the magnitude of weight loss on non-alcoholic fatty liver disease: A systematic review and meta-analysis. Metabolism. 2021 Feb;115:154455. doi: 10.1016/j.metabol.2020.154455. Epub 2020 Nov 29. PMID 33259835
- [Result] Sheka AC, Adeyi O, Thompson J, Hameed B, Crawford PA, Ikramuddin S. Nonalcoholic Steatohepatitis: A Review. JAMA. 2020 Mar 24;323(12):1175-1183. doi: 10.1001/jama.2020.2298. PMID 32207804
- [Result] Hallsworth K, Thoma C, Moore S, Ploetz T, Anstee QM, Taylor R, Day CP, Trenell MI. Non-alcoholic fatty liver disease is associated with higher levels of objectively measured sedentary behaviour and lower levels of physical activity than matched healthy controls. Frontline Gastroenterol. 2015 Jan;6(1):44-51. doi: 10.1136/flgastro-2014-100432. Epub 2014 Jun 30. PMID 25580206
- [Result] Koolhaas CM, van Rooij FJ, Cepeda M, Tiemeier H, Franco OH, Schoufour JD. Physical activity derived from questionnaires and wrist-worn accelerometers: comparability and the role of demographic, lifestyle, and health factors among a population-based sample of older adults. Clin Epidemiol. 2017 Dec 18;10:1-16. doi: 10.2147/CLEP.S147613. eCollection 2018. PMID 29296097
- [Result] Gerber L, Otgonsuren M, Mishra A, Escheik C, Birerdinc A, Stepanova M, Younossi ZM. Non-alcoholic fatty liver disease (NAFLD) is associated with low level of physical activity: a population-based study. Aliment Pharmacol Ther. 2012 Oct;36(8):772-81. doi: 10.1111/apt.12038. Epub 2012 Sep 8. PMID 22958053
- [Result] Joo JH, Kim HJ, Park EC, Jang SI. Association between sitting time and non-alcoholic fatty live disease in South Korean population: a cross-sectional study. Lipids Health Dis. 2020 Sep 23;19(1):212. doi: 10.1186/s12944-020-01385-6. PMID 32967678
- [Result] St George A, Bauman A, Johnston A, Farrell G, Chey T, George J. Independent effects of physical activity in patients with nonalcoholic fatty liver disease. Hepatology. 2009 Jul;50(1):68-76. doi: 10.1002/hep.22940. PMID 19444870
- [Result] Zelber-Sagi S, Nitzan-Kaluski D, Goldsmith R, Webb M, Zvibel I, Goldiner I, Blendis L, Halpern Z, Oren R. Role of leisure-time physical activity in nonalcoholic fatty liver disease: a population-based study. Hepatology. 2008 Dec;48(6):1791-8. doi: 10.1002/hep.22525. PMID 18972405
- [Result] Mansour-Ghanaei R, Mansour-Ghanaei F, Naghipour M, Joukar F. The Lifestyle Characteristics in Non-Alcoholic Fatty Liver Disease in the PERSIAN Guilan Cohort Study. Open Access Maced J Med Sci. 2019 Sep 14;7(19):3313-3318. doi: 10.3889/oamjms.2019.647. eCollection 2019 Oct 15. PMID 31949537
- [Result] Rinella ME, Neuschwander-Tetri BA, Siddiqui MS, Abdelmalek MF, Caldwell S, Barb D, Kleiner DE, Loomba R. AASLD Practice Guidance on the clinical assessment and management of nonalcoholic fatty liver disease. Hepatology. 2023 May 1;77(5):1797-1835. doi: 10.1097/HEP.0000000000000323. Epub 2023 Mar 17. No abstract available. PMID 36727674
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on non-invasive tests for evaluation of liver disease severity and prognosis - 2021 update. J Hepatol. 2021 Sep;75(3):659-689. doi: 10.1016/j.jhep.2021.05.025. Epub 2021 Jun 21. PMID 34166721
- [Result] Maximos M, Bril F, Portillo Sanchez P, Lomonaco R, Orsak B, Biernacki D, Suman A, Weber M, Cusi K. The role of liver fat and insulin resistance as determinants of plasma aminotransferase elevation in nonalcoholic fatty liver disease. Hepatology. 2015 Jan;61(1):153-60. doi: 10.1002/hep.27395. Epub 2014 Nov 25. PMID 25145475
- [Result] Anstee QM, Day CP. The Genetics of Nonalcoholic Fatty Liver Disease: Spotlight on PNPLA3 and TM6SF2. Semin Liver Dis. 2015 Aug;35(3):270-90. doi: 10.1055/s-0035-1562947. Epub 2015 Sep 17. PMID 26378644
- [Result] Krawczyk M, Rau M, Schattenberg JM, Bantel H, Pathil A, Demir M, Kluwe J, Boettler T, Lammert F, Geier A; NAFLD Clinical Study Group. Combined effects of the PNPLA3 rs738409, TM6SF2 rs58542926, and MBOAT7 rs641738 variants on NAFLD severity: a multicenter biopsy-based study. J Lipid Res. 2017 Jan;58(1):247-255. doi: 10.1194/jlr.P067454. Epub 2016 Nov 11. PMID 27836992
- [Result] Akuta N, Kawamura Y, Arase Y, Suzuki F, Sezaki H, Hosaka T, Kobayashi M, Kobayashi M, Saitoh S, Suzuki Y, Ikeda K, Kumada H. Relationships between Genetic Variations of PNPLA3, TM6SF2 and Histological Features of Nonalcoholic Fatty Liver Disease in Japan. Gut Liver. 2016 May 23;10(3):437-45. doi: 10.5009/gnl15163. PMID 26610348
- [Result] Romeo S, Kozlitina J, Xing C, Pertsemlidis A, Cox D, Pennacchio LA, Boerwinkle E, Cohen JC, Hobbs HH. Genetic variation in PNPLA3 confers susceptibility to nonalcoholic fatty liver disease. Nat Genet. 2008 Dec;40(12):1461-5. doi: 10.1038/ng.257. Epub 2008 Sep 25. PMID 18820647
- [Result] Trepo E, Romeo S, Zucman-Rossi J, Nahon P. PNPLA3 gene in liver diseases. J Hepatol. 2016 Aug;65(2):399-412. doi: 10.1016/j.jhep.2016.03.011. Epub 2016 Mar 30. PMID 27038645
- [Result] Boeckmans J, Gatzios A, Schattenberg JM, Koek GH, Rodrigues RM, Vanhaecke T. PNPLA3 I148M and response to treatment for hepatic steatosis: A systematic review. Liver Int. 2023 May;43(5):975-988. doi: 10.1111/liv.15533. Epub 2023 Feb 16. PMID 36719059
- [Result] Stens NA, Bakker EA, Manas A, Buffart LM, Ortega FB, Lee DC, Thompson PD, Thijssen DHJ, Eijsvogels TMH. Relationship of Daily Step Counts to All-Cause Mortality and Cardiovascular Events. J Am Coll Cardiol. 2023 Oct 10;82(15):1483-1494. doi: 10.1016/j.jacc.2023.07.029. Epub 2023 Sep 6. PMID 37676198
- [Result] Schneider CV, Zandvakili I, Thaiss CA, Schneider KM. Physical activity is associated with reduced risk of liver disease in the prospective UK Biobank cohort. JHEP Rep. 2021 Mar 2;3(3):100263. doi: 10.1016/j.jhepr.2021.100263. eCollection 2021 Jun. PMID 33898961